CLINICAL TRIAL: NCT01401647
Title: Amiodarone, Lidocaine or Neither for Out-Of-Hospital Cardiac Arrest Due to Ventricular Fibrillation (VF) or Ventricular Tachycardia (VT)
Brief Title: Amiodarone, Lidocaine or Neither for Out-Of-Hospital Cardiac Arrest Due to Ventricular Fibrillation or Tachycardia
Acronym: ALPS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Canadian Institutes of Health Research (CIHR) (Other Government); Heart and Stroke Foundation of Canada (Other); American Heart Association (Other); Defence Research and Development Canada (Industry); U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, Susanne May, Associate Professor, Biostatistics, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 40605-D; 5U01HL077863-07 (NIH)
Record Dates: First submitted 2011-07-08; First posted 2011-07-25 (Estimated); Results first posted 2017-01-30 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; cardiopulmonary resuscitation; ventricular fibrillation; pulseless ventricular tachycardia; Non-traumatic Out of Hospital Cardiac Arrest (OOHCA)
MeSH Terms: conditions — Heart Arrest; Ventricular Fibrillation | interventions — Amiodarone; Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Amiodarone (Active Comparator): Intravenous (IV) or intraosseous (IO) administration of amiodarone if VF/pulseless VT reoccurs after initial defibrillation.
  Interventions: Drug: amiodarone
- Lidocaine (Active Comparator): IV or IO administration of lidocaine if VF/pulseless VT reoccurs after initial defibrillation.
  Interventions: Drug: Lidocaine
- Normal saline (Placebo Comparator): IV or IO administration of normal saline if VF/pulseless VT reoccurs after initial defibrillation.
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: amiodarone — 300 mg will be given IV/IO push for reoccurrence of ventricular fibrillation or pulseless ventricular tachycardia after 1 or more shocks. A second dose of 150 mg will be given if VF/pulseless VT reoccurs after initial dose and a subsequent shock. The initial dose for patients estimated to be less than 100 pounds will be 150 mg, followed by a second dose of 150 mg if the VF/pulseless VT persists.
  Other Names: PM 101, Nexterone
  Arms: Amiodarone
Drug: Lidocaine — 120 mg will be given IV/IO push with reoccurrence of ventricular fibrillation or pulseless ventricular tachycardia after 1 or more shocks. A second dose of 60 mg will be given if VF/pulseless VT reoccurs after initial dose and a subsequent shock. The initial dose for patients estimated to be less than 100 pounds will be 60 mg, followed by a second dose of 60 mg if the VF/pulseless VT persists.
  Other Names: lidocaine hydrochloride
  Arms: Lidocaine
Other: Normal saline — 6 cc of normal saline (NS) will be given IV/IO push for reoccurrence of ventricular fibrillation or pulseless ventricular tachycardia after 1 or more shocks. A second dose of 3 cc will be given if VF/pulseless VT reoccurs after initial dose and a subsequent shock. The initial dose for patients estimated to be less than 100 pounds will be 3 cc, followed by a second dose of 3 cc if the VF/pulseless VT persists.
  Arms: Normal saline

SUMMARY:
The primary objective of the trial is to determine if survival to hospital discharge is improved with early therapeutic administration of a new Captisol-Enabled formulation of IV amiodarone (Nexterone-PM101) compared to placebo.

DETAILED DESCRIPTION:
The primary objective of the trial is to determine if survival to hospital discharge is improved with early therapeutic administration of a new Captisol-Enabled formulation of IV amiodarone (PM101) compared to placebo.

The corresponding null hypothesis is that survival to hospital discharge is identically distributed when out-of-hospital VF/VT arrest is treated with PM101 or placebo.

The secondary objectives of the trial are to determine if survival to hospital discharge is improved with early therapeutic administration of:

1. Lidocaine compared to placebo
2. PM101 compared to lidocaine The corresponding null hypotheses are that survival to hospital admission is identically distributed when out-of-hospital VF/VT arrest is treated with lidocaine as compared with placebo, and with PM101 as compared with lidocaine.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years or local age of consent
* Non-traumatic out-of-hospital cardiac arrest treated by Resuscitation Outcomes Consortium (ROC) emergency medical services (EMS) with advanced life support capability
* VF or pulseless VT presenting as the initial arrest arrhythmia or results from conversion of another arrhythmia (such as transient asystole or pulseless electrical activity)
* Incessant or recurrent VF/VT after receipt of ≥ 1 shocks
* Established vascular access

Exclusion Criteria:

* Asystole or pulseless electrical activity (PEA) as the initial arrest rhythm who never transition to VF or pulseless VT
* Written advance directive to not attempt resuscitation (DNAR)
* Blunt, penetrating, or burn-related injury
* Exsanguination
* Protected populations (prisoners, pregnancy, children under local age of consent)
* Treated exclusively by non-ROC EMS agency/provider, or by basic life support-only capable ROC EMS providers
* Prior receipt of open label lidocaine or amiodarone during resuscitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3024 (Actual)
Dates: Start 2012-05; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myron Weisfeldt, MD, Study Chair — Johns Hopkins University
Locations (9):
- United States (7):
  - Alabama Resuscitation Center, Birmingham, Alabama
  - UCSD-San Diego Resuscitation Center, San Diego, California
  - Portland Resuscitation Outcomes Consortium, Oregon Health & Sciences University, Portland, Oregon
  - The Pittsburgh Resuscitation Network, University of Pittsburgh, Pittsburgh, Pennsylvania
  - Dallas Center for Resuscitation Research, University of Texas Southwestern Medical Center, Dallas, Texas
  - Seattle-King County Center for Resuscitation Research, University of Washington, Seattle, Washington
  - Milwaukee Resuscitation Network, Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - University of Ottawa/University of British Columbia Collaborative RCC, Ottawa Health Research, Ottawa, Ontario
  - Toronto Regional Resuscitation Research Out-of-Hospital Network, University of Toronto, Toronto, Ontario

REFERENCES:
- [Derived] Kudenchuk PJ, Leroux BG, Daya M, Rea T, Vaillancourt C, Morrison LJ, Callaway CW, Christenson J, Ornato JP, Dunford JV, Wittwer L, Weisfeldt ML, Aufderheide TP, Vilke GM, Idris AH, Stiell IG, Colella MR, Kayea T, Egan D, Desvigne-Nickens P, Gray P, Gray R, Straight R, Dorian P; Resuscitation Outcomes Consortium Investigators. Antiarrhythmic Drugs for Nonshockable-Turned-Shockable Out-of-Hospital Cardiac Arrest: The ALPS Study (Amiodarone, Lidocaine, or Placebo). Circulation. 2017 Nov 28;136(22):2119-2131. doi: 10.1161/CIRCULATIONAHA.117.028624. Epub 2017 Sep 13. PMID 28904070
- [Derived] Kudenchuk PJ, Brown SP, Daya M, Rea T, Nichol G, Morrison LJ, Leroux B, Vaillancourt C, Wittwer L, Callaway CW, Christenson J, Egan D, Ornato JP, Weisfeldt ML, Stiell IG, Idris AH, Aufderheide TP, Dunford JV, Colella MR, Vilke GM, Brienza AM, Desvigne-Nickens P, Gray PC, Gray R, Seals N, Straight R, Dorian P; Resuscitation Outcomes Consortium Investigators. Amiodarone, Lidocaine, or Placebo in Out-of-Hospital Cardiac Arrest. N Engl J Med. 2016 May 5;374(18):1711-22. doi: 10.1056/NEJMoa1514204. Epub 2016 Apr 4. PMID 27043165
- See also: ROC Public Homepage — http://roc.uwctc.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Amiodarone | Lidocaine | Normal Saline
Started | 972 | 993 | 1059
Completed | 968 | 985 | 1056
Not Completed | 4 | 8 | 3
Not completed — Withdrawal by Subject | 1 | 5 | 2
Not completed — Lost to Follow-up | 3 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amiodarone | Lidocaine | Normal Saline | Total
Number analyzed (Participants) | 972 | 993 | 1059 | 3024
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (14.0) | 63.4 (14.7) | 63.1 (14.6) | 63.5 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 211 | 177 | 215 | 603
  Male | 761 | 816 | 844 | 2421
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 2 | 4 | 10
  Asian | 18 | 17 | 25 | 60
  Native Hawaiian or Other Pacific Islander | 3 | 4 | 5 | 12
  Black or African American | 95 | 96 | 97 | 288
  White | 334 | 315 | 340 | 989
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 518 | 559 | 587 | 1664

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Survive From the Time of Cardiac Arrest to Hospital Discharge
Description: Patients may die in the field (outside of the hospital at the time of the cardiac arrest), at the emergency room, in the hospital, or they are discharged alive from the hospital.
Time Frame: Patients will be followed from the time of the cardiac arrest until death, hospital discharge, or December 31, 2015, whichever occurs first.
Population: The primary objective is to determine if survival to hospital discharge is improved with early therapeutic administration of IV amiodarone (PM101) compared to placebo.The secondary objectives of the trial are to determine if survival to hospital discharge is improved with early therapeutic administration of Lidocaine vs placebo; PM101 vs lidocaine.
Measure: Number; unit: participants
Arm/Group | Amiodarone | Lidocaine | Normal Saline
Number analyzed (Participants) | 968 | 985 | 1056
participants | 237 | 233 | 222

2. Secondary Outcome: Number of Participants Scoring at or Below a 3 on the MRS Scale
Description: Neurologic status at discharge will be assessed using the modified Rankin Score (MRS). A higher value indicates a worse outcome. 0-No symptoms at all; 1-No significant disability despite symptoms; able to carry out all usual duties and activities, 2-Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance, 3-Moderate disability; requiring some help, but able to walk without assistance; 4-Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance, 5-Severe disability; bedridden, incontinent and requiring constant nursing care and attention; 6-Dead
Time Frame: as for outcome 1
Population: MRS as a secondary outcome is not available on all patients that we have survival for.
Measure: Count of Participants; unit: Participants
Arm/Group | Amiodarone | Lidocaine | Normal Saline
Number analyzed (Participants) | 965 | 984 | 1055
Participants | 182 | 172 | 175

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time a participating agency arrived on scene and up to 24 hours after Emergency Department arrival this results in adverse events reporting for up to 2 days.
Description: The following are commonly observed in patients who experience cardiac arrest or resuscitative efforts, and may or may not be attributable to specific resuscitation therapies. These were monitored and reported but not considered as adverse events of the study intervention. These include, but not limited to: pulmonary edema, airway bleeding, death, Clinical diagnoses of pneumonia, sepsis, cerebral bleeding, stroke, seizures, rearrest, serious rib fractures, and sternal fractures.
Arm/Group | Amiodarone | Lidocaine | Normal Saline
Serious Adverse Events (participants affected / at risk) | 0/972 | 0/993 | 0/1059
Other Adverse Events (participants affected / at risk) | 515/972 | 548/993 | 476/1059
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Amiodarone (N=972) | Lidocaine (N=993) | Normal Saline (N=1059)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 202 | 209 | 184
Hypotension requiring vasopressors (Cardiac disorders) | 118 | 114 | 102
Rearrest (Cardiac disorders) | 57 | 76 | 60
Seizures or potential seizures (Nervous system disorders) | 35 | 49 | 32
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 103 | 100 | 98

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days